CLINICAL TRIAL: NCT06747247
Title: A Double-blind, Randomized, Placebo-controlled, Single-dose Escalation and Multi-dose Escalation Clinical Study Evaluating the Safety, Tolerability, and Efficacy of MT1013 in Hemodialysis Subjects With Secondary Hyperparathyroidism, Along With a Single-arm Study Assessing the Long-term Efficacy and Safety of MT1013
Brief Title: A Clinical Study Evaluating the Safety, Tolerability, and Efficacy of MT1013 in Hemodialysis Subjects With Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT1013-II-C01
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Secondary Hyperparathyroidism (SHPT) in Subjects With Chronic Kidney Disease (CKD) on Hemodialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Intervention Model Description: This study consists of the following three cohorts:
  SAD Cohort: All subjects will receive a single dose only after a single hemodialysis session and will be followed up on Day 8±1.
  MAD Cohort: All subjects will undergo regular hemodialysis three times per week. Dosing will occur once after each hemodialysis session, continuing for either 2 or 4 weeks (treatment period). Subjects will undergo safety follow-up on Day 16+2 or 30+2 and Day 21±2 or 35±2.
  Long-term Dosing Cohort: All subjects will undergo hemodialysis three times per week. Dosing will occur once after each hemodialysis session and will continue for 52 weeks. The first 10 weeks constitute the dose titration period, during which the drug dose is titrated every 3 weeks based on iPTH and serum corrected calcium levels. During other treatment periods, the drug dose may be adjusted based on iPTH and serum corrected calcium levels.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- MT1013 for SAD (Experimental): Single ascending doses of MT1013
  Interventions: Drug: Single ascending doses of MT1013
- Placebo for SAD (Placebo Comparator): Placebo comparator for SAD
  Interventions: Drug: Single ascending doses of MT1013
- MT1013 for MAD (Experimental): Multiple ascending doses of MT1013
  Interventions: Drug: Multiple ascending doses of MT1013
- Placebo for MAD (Placebo Comparator): Placebo comparator for MAD
  Interventions: Drug: Multiple ascending doses of MT1013
- Long-term Dosing Cohort (Experimental): Dose titration period covers the first 10 weeks , followed by maintenance dosing period, for a total treatment duration of 52 weeks
  Interventions: Drug: Long-term Dosing Cohort

INTERVENTIONS:
Drug: Long-term Dosing Cohort — All subjects will undergo regular hemodialysis three times per week. Administration of MT1013occurs once after each hemodialysis session and will continue for 52 weeks. The first 10 weeks constitute the dose-titration period, during which the drug dose is titrated every 3 weeks based on iPTH and serum corrected calcium levels.
  During the maintenance dosing period, doses is adjusted based on iPTH and serum corrected calcium levels.
  Arms: Long-term Dosing Cohort
Drug: Single ascending doses of MT1013 — All subjects will receive a single dose (MT1013 or placebo) only after a single hemodialysis session
  Arms: MT1013 for SAD; Placebo for SAD
Drug: Multiple ascending doses of MT1013 — All subjects will undergo hemodialysis three times per week. Dosing (MT1013 or placebo) will occur once after each hemodialysis session, continuing for either 2 or 4 weeks (treatment period).
  Arms: MT1013 for MAD; Placebo for MAD

SUMMARY:
A multicenter, Phase II, randomized, double-blind, single ascending dose (SAD) and multiple ascending dose (MAD), as well as single-arm clinical study evaluating the long-term efficacy and safety of MT1013 in hemodialysis subjects with secondary hyperparathyroidism. The SAD study consists of five cohorts at doses of 5, 10, 20, 40, and 60 mg. The MAD study consists of three cohorts at doses of 5, 10, and 20 mg. In both the SAD and MAD studies, each cohort includes 8 subjects (6 subjects receive the active investigational drug, and 2 subjects receive matching placebo), and the cohorts are conducted sequentially. In the long-term dosing cohort, all subjects will undergo regular hemodialysis three times per week, receiving the drug once after each hemodialysis session for a total duration of 52 weeks

ELIGIBILITY:
Inclusion Criteria (Subjects must meet all of the following criteria to participate in the trial):

1. Male or non- pregnant, non-lactating female aged 18 to 80;
2. The patient has been on stable, adequate hemodialysis treatment for >3 months prior to screening;
3. Intact parathyroid hormone (iPTH) level of at least 300 pg/mL;
4. Serum calcium (corrected serum calcium if albumin <40 g/L) ≥2.25 mmol/L (9.0mg/dL);
5. Hemoglobin ≥ 8.0 g/dL;
6. Subject is clinically stable, as judged by medical history, physical examination, and routine laboratory tests, apart from chronic renal failure;
7. Able to understand and willing to sign the written informed consent form;
8. Women of childbearing potential must have a negative pregnancy test result prior to enrollment, or be postmenopausal for at least 1 year, or be permanently sterile(i.e., documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) for ≥6 weeks. Fertile men with partners of childbearing potential and women of childbearing potential must use effective contraception (i.e., any combination of two of the following: male or female condom with spermicidal gel,diaphragm, sponge, or cervical cap with spermicidal gel) from signing the informed consent until 90 days after MT1013 infusion.

Postmenopausal is defined as:

Age ≥55 years & amenorrhea for ≥12 months;

Or Age <55 years but no spontaneous menses for at least 2 years;

Or Age <55 years with spontaneous menses within the past 1 year, but currently amenorrheic, and with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels >40 IU/L) or postmenopausal estradiol levels (<5.3 pmol/L or 5 ng/dL) or meeting the laboratory's definition of "postmenopausal range";Having undergone bilateral oophorectomy.

Exclusion Criteria (Subjects meeting any of the following criteria will be excluded from the study):

1 .History of severe ventricular arrhythmia or symptomatic ventricular arrhythmia at screening, or QTc >470 ms for males or >480 ms for females at screening;

2. Subjects with heart failure symptoms，class III or IV by New York Heart Association (NYHA) ， at screening;

3. History of myocardial infarction, coronary angioplasty, or coronary artery bypass graft within the past 6 months;

4. History of seizures or having received treatment for seizures;

5. Prior parathyroidectomy;

6. Serum transaminases (alanine aminotransferase, aspartate aminotransferase) >3 times the upper limit of normal at screening; or serum albumin <30 g/L;

7.History of organ transplant (excluding being on the kidney transplant waiting list), hematopoietic stem cell transplant, or bone marrow transplant; or patients planning to undergo organ transplantation;

8.Severe uncontrolled hypertension, defined as systolic blood pressure >180 mmHg and diastolic blood pressure >100 mmHg despite optimal medical therapy before enrollment;

9.Known malignancy or other comorbidities with a life expectancy of <3 months (except for patients disease-free for ≥5 years, or disease-free for ≥5 years after the last dose of chemotherapy );

10.Known alcohol or illicit drug abuse within 12 months prior to screening, unwillingness or inability to abstain from alcohol for 24 hours prior to each study visit, or unwillingness or inability to limit alcohol consumption to a maximum of 2 drinks per day during the study (one drink is equivalent to 360 mL of regular beer, 150 mL of wine, or 45 mL of 40% alcohol spirits);

11.Positive for human immunodeficiency virus (HIV) or known diagnosis of acquired immunodeficiency syndrome (AIDS) at screening;

12.Subjects positive for hepatitis B surface antigen (HBsAg) at screening (indicative of chronic hepatitis B) AND with serum transaminases (alanine aminotransferase, aspartate aminotransferase) >2 times the upper limit of normal;

13.Positive for hepatitis C virus ribonucleic acid (RNA) by polymerase chain reaction (PCR) at screening (indicative of active hepatitis C - usually screened via hepatitis C antibody [HCV-Ab], with PCR for HCV RNA if HCV-Ab positive);

14.Patients with known hypersensitivity to the investigational product and/or its components;

15.Patients who have participated in another clinical trial and received an investigational drug within 8 weeks prior to the first dose or within 5 half-lives of the investigational drug (whichever is longer);

16. Patients who have previously received MT1013;

17. Subjects who have received cinacalcet treatment within 8 days prior to the first dose;

18. Pregnant or potentially pregnant women or lactating women;

19. Inability to fully comply with the study protocol;

20.Any other medical or psychiatric condition that, in the investigator's opinion, precludes participation in the study;

21. Subjects with active gastrointestinal bleeding or a high risk of astrointestinal bleeding tendency at screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
SAD/MAD :Percentage of treatment-emergent adverse events (TEAEs) | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2
  To investigate the safety and tolerability of MT1013 by assessing the incidence and severity of TEAEs in Single Ascending Dose (SAD Cohort) and Multiple Ascending Doses (MAD Cohort)
Long-term Dosing Cohort: Proportion of subjects with > 30% reduction in serum iPTH compared to baseline level. | 14 weeks
  Proportion of subjects achieving a >30% reduction in serum iPTH from baseline at Week 14.

SECONDARY OUTCOMES:
Change in the mean serum intact parathyroid hormone (iPTH) from baseline | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2. Long-term Dosing Cohort: 52 weeks
  Change in serum intact parathyroid hormone (iPTH) from baseline at each visit
Proportion of subjects achieving a >30% reduction in serum iPTH from baseline | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2. Long-term Dosing Cohort: 52 weeks
  Proportion of subjects achieving a >30% reduction in serum iPTH from baseline at each visit
Change from baseline in corrected Ca | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2. Long-term Dosing Cohort: 52 weeks
  Change in corrected calcium from baseline at each visit
Change from baseline in ionized calcium | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2
  Change in ionized calcium from baseline at each visit
Change in DXA-measured bone mineral density (BMD) at the femoral neck and lumbar spine from baseline | Long-term Dosing Cohort: 52 weeks
  Change in DXA-measured bone mineral density (BMD) at the femoral neck and lumbar spine from baseline at each visit
Incidence and severity of treatment-emergent adverse events (TEAEs) | Long-term Dosing Cohort: 52 weeks
  Incidence and severity of adverse events occurred during the study period
Change from baseline in serum phosphorus | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2
  Change in serum phosphorus from baseline at each visit
Change from baseline in the mean corrected calcium-phosphorus product | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2
  Change in the mean corrected calcium-phosphorus product from baseline at each visit
Assessment change of Bone Turnover Markers - Change from Baseline | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2. Long-term Dosing Cohort: 52 weeks
  Change in PINP from baseline at each visit
Assessment change of Bone Turnover Markers - Change from Baseline | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2. Long-term Dosing Cohort: 52 weeks
  Change in CTX from baseline at each visit
Assessment change of Bone Turnover Markers - Change from Baseline | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2. Long-term Dosing Cohort: 52 weeks
  Change in OC from baseline at each visit
Assessment change of Bone Turnover Markers - Change from Baseline | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2. Long-term Dosing Cohort: 52 weeks
  Change in b-ALP from baseline at each visit
Assessment change of Bone Turnover Markers - Change from Baseline | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2. Long-term Dosing Cohort: 52 weeks
  Change in TRAP-5b from baseline at each visit
Cmax of MT1013 | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2
  Cmax - Maximum plasma concentration
Tmax of MT1013 | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2
  Tmax - Time to reach Cmax
T1/2 of MT1013 | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2
  T1/2 - Elimination half-life
AUC0-tau of MT1013 | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2
  AUC0-tau - Area under the plasma concentration-time curve during one dosing interval
AUC0-t of MT1013 | SAD：on Day 8±1. MAD：on Day 16+2 or 30+2 and Day 21±2 or 35±2
  AUC0-t - Area under the plasma concentration-time curve from time zero to the last measurable concentration

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China